CLINICAL TRIAL: NCT05799313
Title: A Randomized Trial Comparing Home verSus In-office Removal of the percuTaneous Nerve evaluatIon Lead perforMed for the Treatment of Overactive Bladder in Women (STIM Trial)
Brief Title: Home Versus Office Removal of Percutaneous Nerve Evaluation (PNE) Lead
Acronym: STIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-1242
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- At home removal (Experimental)
  Interventions: Other: At home removal
- In office removal (Active Comparator)
  Interventions: Other: In office removal

INTERVENTIONS:
Other: At home removal — Removal of PNE lead at home
  Arms: At home removal
Other: In office removal — Removal of PNE lead in the office
  Arms: In office removal

SUMMARY:
For women undergoing percutaneous nerve evaluation (PNE) for the treatment of overactive bladder the first step is the PNE interstim therapy trial. If the PNE works, patients may opt to have the interstim procedure. The purpose of this study is to see if patients who remove their PNE lead at home have the same satisfaction with the PNE trial as those women who have their lead removed in the office.

DETAILED DESCRIPTION:
Study Identification and Recruitment: Potential subjects will be identified by members of the Center for Urogynecology & Pelvic Reconstructive Surgery at the Cleveland Clinic Main campus, Hillcrest Hospital, Medina Hospital, and Fairview Hospital. Eligible patients who agree to participate will be provided written informed consent administered by the collaborators listed on this IRB. Enrollment and consent will take place either at the time of office consultation prior to the procedure or virtually before the procedure using DocuSign.

Randomization: Randomization will occur prior to PNE placement. Subjects will be randomized to either in-office versus at-home removal of the PNE lead. Randomization will be done according to a computer-generated randomization schedule with the use of the SAS statistical software package (SAS Institute, Cary, NC). Subjects and research personnel will not be blinded to group allocation.

Intervention: PNE will be performed in a standard fashion with the patient placed in a flat prone position. Her lower back will be prepped with antiseptics and she will be draped in sterile fashion. Her coccyx is identified and an area 9cm cephalad to this point will be marked with a pen. A line is then drawn 2 cm bilaterally in a horizontal fashion and points 2 cm cephalad to these points will also be marked to estimate the skin entry point for access into the S3 foramen. Local anesthesia (1% lidocaine) will be infiltrated bilaterally in the marked areas. The PNE kit is opened and the foramen needle is inserted at an approximately 60 degree through one of the marked sites, entering the presumed S3 foramen. The S3 foraminal location is confirmed with any of the following responses: levator ani motor response (perirectal bellows), plantar flexion of the ipsilateral great toe, and/or patient report of perineal sensation. A second foramen needle is then placed on the contralateral side, 4 cm away from the first needle, also at a 60-degree angle, into the S3 foramen. Foraminal location is again confirmed with any of the following responses: levator ani motor response (perirectal bellows), plantar flexion of the ipsilateral great toe, and/or patient report of perineal sensation. Once the S3 foraminal location is confirmed, the stylets are removed and the temporary leads are placed. The leads are tested bilaterally and if similar responses are obtained bilaterally the procedure is complete. The temporary leads are then taped securely to the skin with Tegaderm.

PNE Lead Removal: Patients will complete the trial within 3 to 7 days of the PNE lead being placed.

At Home Removal: Patients will receive a phone call day of removal by study personnel and they will be guided over the phone on how to remove the lead in real time. If there is any question of complete lead removal, they will be asked to upload a picture of their lead to their MyChart or they will text a picture of it to a Cleveland Clinic encrypted mobile phone belonging to one of the study personnel. Confirmation of complete lead removal will be made and documented in the patient's electronic medical record. If there is any concern that the lead was not removed entirely, the patient will be asked to come into the office for a visit and they will bring the removed lead with them.

In Office Removal: The temporary lead will be removed in the office at a scheduled visit by study personnel. Confirmation of complete lead removal will be documented in the patient's electronic medical record.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years of age
* Patients undergoing sacral neuromodulation (SNM) for urinary urgency incontinence or urgency-frequency syndrome

Exclusion Criteria:

* Inability to comprehend written and/or spoken English
* Inability to provide informed consent
* Patients undergoing SNM for other indications (e.g. urinary retention, fecal incontinence,)
* Previous SNM treatment
* No home support to assist with lead removal

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-07 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction between at home versus in office PNE lead removal | 3-7 days
  Patient reported satisfaction on a scale of 0 (not satisfied) to 10 (most satisfied)

SECONDARY OUTCOMES:
Patient percentage of improvement reported in urinary symptoms | 3-7 days
  Patient reported improvement in urinary symptoms on a scale of 0 (least improvement) to 100 (most improvement)
Patient discomfort with PNE trial overall | 3-7 days
  Patient reported discomfort with PNE trial overall on a scale of 0 (no discomfort) to 10 (most discomfort)
Patient discomfort with PNE lead removal | 3-7 days
  Patient reported discomfort with PNE lead removal on a scale of 0 (no discomfort) to 10 (most discomfort)
Patient inconvenience for PNE lead removal | 3-7 days
  Patient reported inconvenience for PNE lead removal on a scale of 0 (not inconvenient) to 10 (most inconvenient)
Patient preference for PNE lead removal at home or in office | 3-7 days
  Patient choice of in office or at home
Physician ease of PNE lead placement | 1 day
  Physician ease of PNE lead placement on a scale of 0 (very difficult) to 10 (very easy)
Patient reported degree of pain of PNE lead placement | 1 day
  Patient reported degree of pain of PNE lead placement on a scale of 0 (no pain) to 10 (most painful)

CONTACTS AND LOCATIONS:
Overall Officials: Cecile A. Ferrando, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No